CLINICAL TRIAL: NCT01018732
Title: A Phase 2b, Open-Label, Multi-Center Study to Evaluate the Persistence of Antibody Response and to Assess the Immune Response to a Booster Dose of MenACWY Conjugate Vaccine in Subjects Previously Vaccinated as Adolescents With Either MenACWY Conjugate Vaccine or Menomune®.
Brief Title: A Study to Evaluate the Persistence and Immune Response to a Booster Dose of MenACWY
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Vaccines (Industry)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: V59P6E1
Record Dates: First submitted 2009-11-18; First posted 2009-11-25 (Estimated); Results first posted 2011-09-13 (Estimated); Last update posted 2015-07-15 (Estimated); Status verified 2015-07

CONDITIONS: Meningococcal Disease; Meningococcal Meningitis
Keywords: Meningococcal; ACWY; Conjugate Vaccine; Meningitis; Adolescents; Persistence
MeSH Terms: conditions — Meningococcal Infections; Meningitis, Meningococcal; Meningitis | interventions — Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- I: MenACWY-CRM vaccine (Experimental): Subjects had been given one dose of Meningococcal ACWY (MenACWY) vaccine conjugated to CRM197 (cross-reactive material-mutant of diptheria toxin) 5 years ago. All subjects were given one dose of the Men ACWY in the present study.
  Interventions: Biological: Novartis Meningococcal (MenACWY-CRM) vaccine
- II: Licensed Polysaccharide Meningococcal vaccine (Experimental): Subjects had been given one dose of a licensed MenACWY polysaccharide meningococcal vaccine (Menomune) 5 years ago. All subjects were given one dose of Men ACWY vaccine in the present study.
  Interventions: Biological: Novartis Meningococcal (MenACWY-CRM) vaccine
- III: Meningococcal Naive (Experimental): Subjects were age matched with groups 1 and 2 (age inclusive: 16 years to 23 years) and enrolled at visit 1 and given one dose of Men ACWY vaccine during the present study.
  Interventions: Biological: Novartis Meningococcal (MenACWY-CRM) vaccine

INTERVENTIONS:
Biological: Novartis Meningococcal (MenACWY-CRM) vaccine — All subjects will have blood draws at Day 1, Day 8, and Day 29.

SUMMARY:
The primary objective is to evaluate the persistence of bactericidal antibodies in adolescent subjects who completed study V59P6 in which they received either Novartis Meningococcal (MenACWY) Conjugate Vaccine or Licensed polysaccharide Men ACWY vaccine (Menomune®). The study will also enroll age-matched subjects who have never received any other meningococcal vaccine (naïve subjects) to serve as an additional control group.

DETAILED DESCRIPTION:
Persistence of antibody response at 5 years after one dose of MenACWY or Menomune

ELIGIBILITY:
Inclusion Criteria:

* Healthy adolescents or adults (age 16-23 years inclusive), either previously enrolled in the parent study or naïve to meningococcal vaccination.
* Female subjects were to be negative for pregnancy

Exclusion Criteria:

* History of meningococcal disease
* Receipt of any meningococcal vaccine outside of parent study (V59P6)
* Serious, acute, or chronic illnesses including HIV infection/disease and any malignancy
* receipt of any vaccine 14 days prior to the study, or expected through the duration of the study
* any condition which in the eyes of the investigator would pose a health risk to the subject or render them inappropriate for a research study

Ages: 16 Years to 23 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 155 (Actual)
Dates: Start 2010-01; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Rochester, Minnesota
  - Pittsburgh, Pennsylvania
  - Seattle, Washington

REFERENCES:
- [Result] Kimura A, Toneatto D, Kleinschmidt A, Wang H, Dull P. Immunogenicity and safety of a multicomponent meningococcal serogroup B vaccine and a quadrivalent meningococcal CRM197 conjugate vaccine against serogroups A, C, W-135, and Y in adults who are at increased risk for occupational exposure to meningococcal isolates. Clin Vaccine Immunol. 2011 Mar;18(3):483-6. doi: 10.1128/CVI.00304-10. Epub 2010 Dec 22. PMID 21177912
- [Result] Jacobson RM, Jackson LA, Reisinger K, Izu A, Odrljin T, Dull PM. Antibody persistence and response to a booster dose of a quadrivalent conjugate vaccine for meningococcal disease in adolescents. Pediatr Infect Dis J. 2013 Apr;32(4):e170-7. doi: 10.1097/INF.0b013e318279ac38. PMID 23114372

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 3 centers in the USA
Pre-assignment Details: All subjects enrolled were included in the trial.
Groups:
- I: MenACWY-CRM Vaccine: Subjects had been given one dose of Meningococcal ACWY (MenACWY)vaccine conjugated to CRM197 (cross-reactive material-mutant of diptheria toxin) 5 years ago
- II: Licensed Polysaccharide Meningococcal Vaccine: Subjects had been given one dose of licensed Meningococcal (Men ACWY) polysaccharide vaccine (Menomune) 5 years ago
- III: Meningococcal Naive: Subjects were between 16 years to 23 years (age-inclusive)and meningococcal vaccine naive
Period: Overall Study
Arm/Group | I: MenACWY-CRM Vaccine | II: Licensed Polysaccharide Meningococcal Vaccine | III: Meningococcal Naive
Started | 50 | 51 | 54
Completed | 49 | 49 | 50
Not Completed | 1 | 2 | 4
Not completed — Lost to Follow-up | 0 | 0 | 3
Not completed — Protocol Violation | 1 | 1 | 0
Not completed — Inappropriate Enrollment | 0 | 1 | 0
Not completed — Unable to Classify | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | I: MenACWY-CRM Vaccine | II: Licensed Polysaccharide Meningococcal Vaccine | III: Meningococcal Naive | Total
Number analyzed (Participants) | 50 | 51 | 54 | 155
Age, Continuous [Mean (Standard Deviation); unit: years] | 18.8 (1.9) | 19.2 (2.0) | 20.5 (2.3) | 19.5 (2.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 28 | 33 | 83
  Male | 28 | 23 | 21 | 72

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Serum Bactericidal Activity >=8 at 5 Years After Primary Vaccination
Description: Persistence of antibody response was measured by the percentage of subjects who showed a serum bactericidal activity with human complement(hSBA) >= 8 [i.e. percentage of subjects with hsBA titer >=8] in previously vaccinated subjects and in age-matched meningococcal vaccine naive subjects. Sera was tested against Neisseria meningitidis serogroups A, C, W-135 and Y
Time Frame: Day 1 (5 years after primary vaccination)
Population: Full analysis set (all subjects who had no major protocol violation as defined prior to database lock).
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- I:MenACWY: Subjects had been given one dose of Meningococcal (MenACWY) vaccine 5 years ago and were given one dose of Men ACWY-CRM vaccine during the study.
- II:Licensed Polysacharide Meningococcal Vaccine: Subjects had been given one dose of licensed polysaccharide meningococcal Serogroup ACWY vaccine(Menomune),5 years ago and were given one dose of Men ACWY-CRM vaccine during the study.
- III: Meningococcal-naive: Subjects were meningococcal vaccine naive and age inclusive (16-23 years)and were given one dose of Men ACWY-CRM vaccine during the study.
Arm/Group | I:MenACWY | II:Licensed Polysacharide Meningococcal Vaccine | III: Meningococcal-naive
Number analyzed (Participants) | 50 | 50 | 53
Percentage of participants
  Men A | 30 [18 to 45] | 44 [30 to 59] | 11 [4 to 23]
  Men C | 76 [62 to 87] | 62 [47 to 75] | 51 [37 to 65]
  Men W-135 | 72 [58 to 84] | 56 [41 to 70] | 51 [37 to 65]
  Men Y | 76 [62 to 87] | 50 [36 to 64] | 55 [40 to 68]

2. Primary Outcome: Geometric Mean Titer After Booster Vaccination
Description: Immunogenicity was measured by serum bactericidal assay with human complement (hSBA) and reported as hSBA Geometric mean titer (GMT) in previously vaccinated subjects and in age-matched meningococcal vaccine-naive subjects. Sera was tested against Neisseria meningitidis serogroups A, C, W-135 and Y
Time Frame: Day 8, Day 29 (5 years after primary vaccination)
Population: Full analysis set
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | I:MenACWY | II:Licensed Polysacharide Meningococcal Vaccine | III: Meningococcal-naive
Number analyzed (Participants) | 49 | 49 | 50
Titer
  Baseline, Men A | 5.16 [3.46 to 7.7] | 7.31 [4.94 to 11] | 3.06 [2.06 to 4.55]
  Day 8, Men A, | 1059 [585 to 1917] | 45 [25 to 80] | 34 [19 to 61]
  Day 29, Men A, (N=48, G I) | 819 [514 to 1305] | 147 [94 to 232] | 113 [72 to 179]
  Baseline, Men C | 20 [13 to 33] | 19 [12 to 31] | 7.34 [4.6 to 12]
  Day 8, Men C | 1603 [893 to 2877] | 36 [20 to 64] | 70 [39 to 124]
  Day 29, Men C | 1217 [717 to 2066] | 51 [30 to 86] | 127 [75 to 214]
  Baseline, Men W-135 | 29 [17 to 49] | 12 [7.02 to 19] | 11 [6.31 to 18]
  Day 8, Men W-135 | 1685 [1042 to 2725] | 34 [21 to 54] | 63 [39 to 101]
  Day 29, Men W-135 | 1644 [1090 to 2481] | 47 [32 to 71] | 79 [52 to 118]
  Baseline, Men Y | 28 [18 to 45] | 7.8 [4.91 to 12] | 8.69 [5.45 to 14]
  Day 8, Men Y, (N=48, GI) | 2561 [1526 to 4298] | 21 [13 to 35] | 64 [39 to 107]
  Day 29, Men Y | 2092 [1340 to 3268] | 63 [41 to 98] | 110 [70 to 170]
Statistical Analysis 1: Comparison: II:Licensed Polysacharide Meningococcal Vaccine vs III: Meningococcal-naive; Day 1, Men A, Pairwise comparison of geometric mean titer; Test type: Superiority or Other; ANOVA; ratio of titer = 2.39, 95% CI 2-sided [1.39 to 4.1]
Statistical Analysis 2: Comparison: I:MenACWY vs II:Licensed Polysacharide Meningococcal Vaccine; Day 1, Men A, Pairwise comparison of geometric mean titer; Test type: Superiority or Other; ANOVA; ratio of titer = 0.71, 95% CI 2-sided [0.42 to 1.2]
Statistical Analysis 3: Comparison: I:MenACWY vs III: Meningococcal-naive; Day 1, Men A, Pairwise comparison of geometric mean titer; Test type: Superiority or Other; ANOVA; ratio of titer = 1.68, 95% CI 2-sided [0.98 to 2.9]
Statistical Analysis 4: Comparison: II:Licensed Polysacharide Meningococcal Vaccine vs III: Meningococcal-naive; Day 8, Men A, Pairwise comparison of geometric mean titer; Test type: Superiority or Other; ANOVA; ratio of titer = 1.31, 95% CI 2-sided [0.59 to 2.91]
Statistical Analysis 5: Comparison: I:MenACWY vs II:Licensed Polysacharide Meningococcal Vaccine; Day 8, Men A, Pairwise comparison of geometric mean titer; Test type: Superiority or Other; ANOVA; ratio of titer = 24, 95% CI 2-sided [11 to 52]
Statistical Analysis 6: Comparison: I:MenACWY vs III: Meningococcal-naive; Day 8, Men A, Pairwise comparison of geometric mean titer; Test type: Superiority or Other; ANOVA; ratio of titer = 31, 95% CI 2-sided [14 to 69]
Statistical Analysis 7: Comparison: II:Licensed Polysacharide Meningococcal Vaccine vs III: Meningococcal-naive; Day 29, Men A, Pairwise comparison of geometric mean titer; Test type: Superiority or Other; ANOVA; ratio of titer = 1.3, 95% CI 2-sided [0.7 to 2.42]
Statistical Analysis 8: Comparison: I:MenACWY vs II:Licensed Polysacharide Meningococcal Vaccine; Day 29, Men A, Pairwise comparison of geometric mean titer; Test type: Superiority or Other; ANOVA; ratio of titer = 5.56, 95% CI 2-sided [3.01 to 10]
Statistical Analysis 9: Comparison: I:MenACWY vs III: Meningococcal-naive; Day 29, Men A, Pairwise comparison of geometric mean titer; Test type: Superiority or Other; ANOVA; ratio of titer = 7.22, 95% CI 2-sided [3.86 to 13]
Statistical Analysis 10: Comparison: II:Licensed Polysacharide Meningococcal Vaccine vs III: Meningococcal-naive; Day 1, Men C, Pairwise comparison of geometric mean titer; Test type: Superiority or Other; ANOVA; ratio of titer = 2.64, 95% CI 2-sided [1.4 to 4.99]
Statistical Analysis 11: Comparison: I:MenACWY vs II:Licensed Polysacharide Meningococcal Vaccine; Day 1, Men C, Pairwise comparison of geometric mean titer; Test type: Superiority or Other; ANOVA; ratio of titer = 1.05, 95% CI 2-sided [0.56 to 1.97]
Statistical Analysis 12: Comparison: I:MenACWY vs III: Meningococcal-naive; Day 1, Men C, Pairwise comparison of geometric mean titer; Test type: Superiority or Other; ANOVA; ratio of titer = 2.78, 95% CI 2-sided [1.47 to 5.27]
Statistical Analysis 13: Comparison: II:Licensed Polysacharide Meningococcal Vaccine vs III: Meningococcal-naive; Day 8, Men C, Pairwise comparison of geometric mean titer; Test type: Superiority or Other; ANOVA; ratio of titer = 0.52, 95% CI 2-sided [0.23 to 1.13]
Statistical Analysis 14: Comparison: I:MenACWY vs II:Licensed Polysacharide Meningococcal Vaccine; Day 8, Men C, Pairwise comparison of geometric mean titer; Test type: Superiority or Other; ANOVA; ratio of titer = 45, 95% CI 2-sided [21 to 97]
Statistical Analysis 15: Comparison: I:MenACWY vs III: Meningococcal-naive; Day 8, Men C, Pairwise comparison of geometric mean titer; Test type: Superiority or Other; ANOVA; ratio of titer = 23, 95% CI 2-sided [10 to 51]
Statistical Analysis 16: Comparison: II:Licensed Polysacharide Meningococcal Vaccine vs III: Meningococcal-naive; Day 29, Men C, Pairwise comparison of geometric mean titer; Test type: Superiority or Other; ANOVA; ratio of titer = 0.4, 95% CI 2-sided [0.2 to 0.82]
Statistical Analysis 17: Comparison: I:MenACWY vs II:Licensed Polysacharide Meningococcal Vaccine; Day 29, Men C, Pairwise comparison of geometric mean titer; Test type: Superiority or Other; ANOVA; ratio of titer = 24, 95% CI 2-sided [12 to 48]
Statistical Analysis 18: Comparison: I:MenACWY vs III: Meningococcal-naive; Day 29, Men C, Pairwise comparison of geometric mean titer; Test type: Superiority or Other; ANOVA; ratio of titer = 9.61, 95% CI 2-sided [4.69 to 20]
Statistical Analysis 19: Comparison: II:Licensed Polysacharide Meningococcal Vaccine vs III: Meningococcal-naive; Day 1, Men W-135, Pairwise comparison of geometric mean titer; Test type: Superiority or Other; ANOVA; ratio of titer = 1.11, 95% CI 2-sided [0.55 to 2.21]
Statistical Analysis 20: Comparison: I:MenACWY vs II:Licensed Polysacharide Meningococcal Vaccine; Day 1, Men W-135, Pairwise comparison of geometric mean titer; Test type: Superiority or Other; ANOVA; ratio of titer = 2.51, 95% CI 2-sided [1.27 to 4.96]
Statistical Analysis 21: Comparison: I:MenACWY vs III: Meningococcal-naive; Day 1, Men W-135, Pairwise comparison of geometric mean titer; Test type: Superiority or Other; ANOVA; ratio of titer = 2.77, 95% CI 2-sided [1.38 to 5.57]
Statistical Analysis 22: Comparison: II:Licensed Polysacharide Meningococcal Vaccine vs III: Meningococcal-naive; Day 8, Men W-135, Pairwise comparison of geometric mean titer; Test type: Superiority or Other; ANOVA; ratio of titer = 0.54, 95% CI 2-sided [0.28 to 1.04]
Statistical Analysis 23: Comparison: I:MenACWY vs II:Licensed Polysacharide Meningococcal Vaccine; Day 8, Men W-135, Pairwise comparison of geometric mean titer; Test type: Superiority or Other; ANOVA; ratio of titer = 50, 95% CI 2-sided [26 to 94]
Statistical Analysis 24: Comparison: I:MenACWY vs III: Meningococcal-naive; Day 8, Men W-135, Pairwise comparison of geometric mean titer; Test type: Superiority or Other; ANOVA; ratio of titer = 27, 95% CI 2-sided [14 to 52]
Statistical Analysis 25: Comparison: II:Licensed Polysacharide Meningococcal Vaccine vs III: Meningococcal-naive; Day 29, Men W-135, Pairwise comparison of geometric mean titer; Test type: Superiority or Other; ANOVA; ratio of titer = 0.6, 95% CI 2-sided [0.34 to 1.04]
Statistical Analysis 26: Comparison: I:MenACWY vs II:Licensed Polysacharide Meningococcal Vaccine; Day 29, Men W-135, Pairwise comparison of geometric mean titer; Test type: Superiority or Other; ANOVA; ratio of titer = 35, 95% CI 2-sided [20 to 60]
Statistical Analysis 27: Comparison: I:MenACWY vs III: Meningococcal-naive; Day 29, Men W-135, Pairwise comparison of geometric mean titer; Test type: Superiority or Other; ANOVA; ratio of titer = 21, 95% CI 2-sided [12 to 36]
Statistical Analysis 28: Comparison: II:Licensed Polysacharide Meningococcal Vaccine vs III: Meningococcal-naive; Day 1, Men Y, Pairwise comparison of geometric mean titer; Test type: Superiority or Other; ANOVA; ratio of titer = 0.9, 95% CI 2-sided [0.48 to 1.69]
Statistical Analysis 29: Comparison: I:MenACWY vs II:Licensed Polysacharide Meningococcal Vaccine; Day 1, Men Y, Pairwise comparison of geometric mean titer; Test type: Superiority or Other; ratio of titer = 3.61, 95% CI 2-sided [1.94 to 6.74]
Statistical Analysis 30: Comparison: I:MenACWY vs III: Meningococcal-naive; Day 1, Men Y, Pairwise comparison of geometric mean titer; Test type: Superiority or Other; ANOVA; ratio of titer = 3.24, 95% CI 2-sided [1.71 to 6.13]
Statistical Analysis 31: Comparison: II:Licensed Polysacharide Meningococcal Vaccine vs III: Meningococcal-naive; Day 8, Men Y, Pairwise comparison of geometric mean titer; Test type: Superiority or Other; ANOVA; ratio of titer = 0.33, 95% CI 2-sided [0.16 to 0.66]
Statistical Analysis 32: Comparison: I:MenACWY vs II:Licensed Polysacharide Meningococcal Vaccine; Day 8, Men Y, Pairwise comparison of geometric mean titer; Test type: Superiority or Other; ANOVA; ratio of titer = 121, 95% CI 2-sided [61 to 241]
Statistical Analysis 33: Comparison: I:MenACWY vs III: Meningococcal-naive; Day 8, Men Y, Pairwise comparison of geometric mean titer; Test type: Superiority or Other; ANOVA; ratio of titer = 40, 95% CI 2-sided [20 to 80]
Statistical Analysis 34: Comparison: II:Licensed Polysacharide Meningococcal Vaccine vs III: Meningococcal-naive; Day 29, Men Y, Pairwise comparison of geometric mean titer; Test type: Superiority or Other; ANOVA; ratio of titer = 0.58, 95% CI 2-sided [0.32 to 1.05]
Statistical Analysis 35: Comparison: I:MenACWY vs II:Licensed Polysacharide Meningococcal Vaccine; Day 29, Men Y, Pairwise comparison of geometric mean titer; Test type: Superiority or Other; ANOVA; ratio of titer = 33, 95% CI 2-sided [18 to 60]
Statistical Analysis 36: Comparison: I:MenACWY vs III: Meningococcal-naive; Day 29, Men Y, Pairwise comparison of geometric mean titer; Test type: Superiority or Other; ANOVA; ratio of titer = 19, 95% CI 2-sided [10 to 35]

3. Secondary Outcome: Percentage of Participants With Serum Bactericidal Activity >=4 at 5 Years After Primary Vaccination
Description: Persistence was measured by percentage of subjects with serum bactericidal activity with human complement (hSBA) >= 4 in previously vaccinated subjects and in age-matched meningococcal vaccine naive subjects. Sera was tested against Neisseria meningitidis serogroups A, C, W-135 and Y
Time Frame: Day 1 (5 years after primary vaccination )
Population: Full analysis set
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | I:MenACWY | II:Licensed Polysacharide Meningococcal Vaccine | III: Meningococcal-naive
Number analyzed (Participants) | 50 | 50 | 53
Percentage of participants
  Men A | 34 [21 to 49] | 50 [36 to 64] | 23 [12 to 36]
  Men C | 84 [71 to 93] | 68 [53 to 80] | 70 [56 to 82]
  Men W-135 | 80 [66 to 90] | 58 [43 to 72] | 55 [40 to 68]
  Men Y | 76 [62 to 87] | 60 [45 to 74] | 60 [46 to 74]

4. Secondary Outcome: Geometric Mean Titer at 5 Years After Primary Vaccination
Description: Persistence was measured by serum bactericidal assay with human complement(hSBA) and expressed as hSBA GMT in previously vaccinated subjects and in age-matched meningococcal vaccine naive subjects. Sera was tested against Neisseria meningitidis serogroups A, C, W-135 and Y
Time Frame: Day 1 (5 years after primary vaccination )
Population: Full analysis set
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | I:MenACWY | II:Licensed Polysacharide Meningococcal Vaccine | III: Meningococcal-naive
Number analyzed (Participants) | 50 | 50 | 53
Titer
  Men A | 5.21 [3.51 to 7.74] | 7.56 [5.12 to 11] | 3 [2.05 to 4.4]
  Men C | 20 [12 to 31] | 19 [12 to 30] | 7.62 [4.86 to 12]
  Men W-135 | 28 [17 to 46] | 12 [7.17 to 20] | 11 [6.53 to 17]
  Men Y | 27 [17 to 43] | 7.67 [4.85 to 12] | 9.38 [5.98 to 15]

5. Secondary Outcome: Percentage of Participants With Serum Bactericidal Activity >=4 After Booster Vaccination
Description: Immunogenicity was measured by serum bactericidal assay with human complement (hSBA) >= 4 in previously vaccinated subjects and in age-matched meningococcal vaccine naive subjects. Sera was tested against Neisseria meningitidis serogroups A, C, W-135 and Y.
Time Frame: Day 7, Day 28 post booster (5 years after primary vaccination)
Population: Full Analysis set
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | I:MenACWY | II:Licensed Polysacharide Meningococcal Vaccine | III: Meningococcal-naive
Number analyzed (Participants) | 49 | 49 | 50
Percentage of participants
  Day 7 post booster, Men A | 100 [93 to 100] | 76 [61 to 87] | 66 [51 to 79]
  Day 28 post booster, Men A | 98 [89 to 100] | 94 [83 to 99] | 92 [81 to 98]
  Day 7 post booster, Men C | 100 [93 to 100] | 82 [68 to 91] | 94 [83 to 99]
  Day 28 post booster, Men C | 100 [93 to 100] | 90 [78 to 97] | 98 [89 to 100]
  Day 7 post booster, Men W-135 | 100 [93 to 100] | 86 [73 to 94] | 92 [81 to 98]
  Day 28 post booster, Men W-135 | 100 [93 to 100] | 94 [83 to 99] | 94 [83 to 99]
  Day 7 post booster, Men Y | 98 [89 to 100] | 78 [63 to 88] | 92 [81 to 98]
  Day 28 post booster, Men Y | 100 [93 to 100] | 100 [93 to 100] | 100 [93 to 100]

6. Secondary Outcome: Percentage of Participants With Serum Bactericidal Activity >=8 After Booster Vaccination
Description: Immunogenicity was measured by serum bactericidal assay with human complement (hSBA) >= 8 in previously vaccinated subjects and in age-matched meningococcal vaccine naive subjects. Sera was tested against Neisseria meningitidis serogroups A, C, W-135 and Y.
Time Frame: Day 7, Day 28 post booster (5 years after primary vaccination)
Population: Full Analysis set
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | I:MenACWY | II:Licensed Polysacharide Meningococcal Vaccine | III: Meningococcal-naive
Number analyzed (Participants) | 49 | 49 | 50
Percentage of participants
  Day 7 post booster, Men A | 100 [93 to 100] | 73 [59 to 85] | 64 [49 to 77]
  Day 28 post booster, Men A | 98 [89 to 100] | 94 [83 to 99] | 92 [81 to 98]
  Day 7 post booster, Men C | 100 [93 to 100] | 78 [63 to 88] | 90 [78 to 97]
  Day 28 post booster, Men C | 100 [93 to 100] | 84 [70 to 93] | 98 [89 to 100]
  Day 7 post booster, Men W-135 | 100 [93 to 100] | 84 [70 to 93] | 88 [76 to 95]
  Day 28 post booster, Men W-135 | 100 [93 to 100] | 92 [80 to 98] | 94 [83 to 99]
  Day 7 post booster, Men Y | 98 [89 to 100] | 76 [61 to 87] | 90 [78 to 97]
  Day 28 post booster, Men Y | 100 [93 to 100] | 96 [86 to 100] | 98 [89 to 100]

7. Secondary Outcome: Geometric Mean Ratio After Booster Vaccination
Description: Ratios are expressed as geometric mean titer at Day 8: Day 1 and at Day 29:Day 1
Time Frame: Day 8 and Day 29 (at 5 Years After Primary Vaccination)
Population: full analysis set
Measure: Mean (95% Confidence Interval); unit: Geometric mean ratio
Arm/Group | I:MenACWY | II:Licensed Polysacharide Meningococcal Vaccine | III: Meningococcal-naive
Number analyzed (Participants) | 49 | 49 | 50
Geometric mean ratio
  Men A (Day 8:1) | 205 [113 to 373] | 6.1 [3.4 to 11] | 11 [6.17 to 20]
  Men A (Day 29:1), N=48, N=49, N=50 | 155 [92 to 262] | 20 [12 to 33] | 37 [22 to 62]
  Men C (Day 8:1) | 78 [47 to 130] | 1.85 [1.13 to 3.03] | 9.48 [5.76 to 16]
  Men C (Day 29:1) | 60 [37 to 97] | 2.64 [1.64 to 4.24] | 17 [11 to 28]
  Men W-135 (Day 8:1) | 58 [34 to 97] | 2.92 [1.75 to 4.87] | 5.95 [3.55 to 9.99]
  Men W-135 (Day 29:1) | 56 [33 to 95] | 4.06 [2.43 to 6.77] | 7.48 [4.46 to 13]
  Men Y (Day 8:1), N=48, N=49, N=50 | 96 [56 to 167] | 2.69 [1.58 to 4.58] | 7.29 [4.26 to 12]
  Men Y (Day 29:1) | 74 [43 to 129] | 8.12 [4.73 to 14] | 13 [7.3 to 22]

8. Secondary Outcome: Percentage of Subjects With hSBA Seroresponse After Booster Vaccination
Description: For a subject with hSBA titer <4 at baseline, seroresponse is defined as a postvaccination hSBA titer >=8; and for a subject with hSBA titer >=4 at baseline, seroresponse is defined as a postvaccination hSBA titer of at least 4 times the baseline. Sera was tested against Neisseria meningitidis serogroups A, C, W-135 and Y.
Time Frame: Day 8, Day 29 (5 years after primary vaccination)
Population: Full analysis set
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | I:MenACWY | II:Licensed Polysacharide Meningococcal Vaccine | III: Meningococcal-naive
Number analyzed (Participants) | 49 | 49 | 50
Percentage of participants
  Men A, Day 8 | 100 [93 to 100] | 51 [36 to 66] | 60 [45 to 74]
  Men A, Day 29 | 100 [93 to 100] | 76 [61 to 87] | 90 [78 to 97]
  Men C, Day 8 | 96 [86 to 100] | 16 [7 to 30] | 62 [47 to 75]
  Men C, Day 29 | 96 [86 to 100] | 31 [18 to 45] | 80 [66 to 90]
  Men W-135, Day 8 | 96 [86 to 100] | 37 [23 to 52] | 48 [34 to 63]
  Men W-135, Day 29 | 98 [89 to 100] | 47 [33 to 62] | 58 [43 to 72]
  Men Y, Day 8, (N=48, G I) | 94 [83 to 99] | 33 [20 to 48] | 54 [39 to 68]
  Men Y, Day 29 | 94 [83 to 99] | 55 [40 to 69] | 76 [62 to 87]

9. Secondary Outcome: Number of Participants With at Least One Reactogenicity Sign After Booster Vaccination
Description: Local and systemic reactions were solicited to assess safety and tolerability of vaccination
Time Frame: Up to Day 7
Measure: Number; unit: participants
Arm/Group | I:MenACWY | II:Licensed Polysacharide Meningococcal Vaccine | III: Meningococcal-naive
Number analyzed (Participants) | 50 | 50 | 53
participants
  Local Reactions (any-total) | 30 | 32 | 40
  Pain (any) | 29 | 27 | 33
  Erythema (any) | 8 | 8 | 15
  Induration (any) | 5 | 8 | 5
  Sytemic Reactions (any-total) | 31 | 25 | 38
  Chills (any) | 7 | 5 | 3
  Nausea (any) | 8 | 9 | 11
  Malaise (any) | 10 | 11 | 15
  Myalgia (any) | 16 | 13 | 17
  Arthalgia (any) | 3 | 5 | 6
  Headache (any) | 21 | 17 | 31
  Fever >= 38C | 0 | 0 | 1
  Stayed at home | 0 | 2 | 2
  Analgesic antipyretic medication used | 10 | 8 | 9

ADVERSE EVENTS:
Time Frame: safety was assessed up to 28 days after vaccination.
Description: All the AEs reported were solicited post-injection reactions
Arm/Group | I: MenACWY-CRM Vaccine | II: Licensed Polysaccharide Meningococcal Vaccine | III: Meningococcal Naive
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50 | 0/53
Other Adverse Events (participants affected / at risk) | 38/50 | 36/50 | 46/53
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | I: MenACWY-CRM Vaccine (N=50) | II: Licensed Polysaccharide Meningococcal Vaccine (N=50) | III: Meningococcal Naive (N=53)
Nausea (Gastrointestinal disorders) | 8 (8) | 9 (9) | 11 (11)
Chills (General disorders) | 7 (7) | 5 (5) | 3 (3)
Injection site erythema (General disorders) | 8 (8) | 8 (8) | 15 (15)
Injection site induration (General disorders) | 5 (5) | 8 (8) | 5 (5)
Injection site pain (General disorders) | 29 (29) | 27 (27) | 33 (33)
Malaise (General disorders) | 10 (10) | 11 (11) | 15 (15)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 5 (5) | 6 (6)
Myalgia (Musculoskeletal and connective tissue disorders) | 18 (18) | 13 (13) | 18 (18)
Headache (Nervous system disorders) | 21 (21) | 17 (17) | 31 (31)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days